CLINICAL TRIAL: NCT04729374
Title: Longidutinal, Dynamic Analysis of COVID-19 Vaccine Induced Adaptive Immune Responses
Brief Title: COVID-19 Vaccine Induced Adaptive Immune Responses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Chao Wu, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: NJGLVAC-001
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV-2; Vaccine; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood (serum, plasma, and DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The coronavirus disease 2019 (COVID-19) caused by the infection of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)，resulting in more than 82 million confirmed cases and caused around 1.8 million deaths, as of 2 January 2021. The ongoing pandemic still poses unprecedented global threat to public health system worldwide. On December 31, 2020, the joint prevention and control agency of China Council announced that Sinopharm SARS-CoV-2 inactivated vaccine had been conditionally approved by National Medical Products Administration, and the protection rate was 79.34%. So far, more than 198 vaccines were currently in preclinical or clinical development. The investigators aimed to initiate an observational cohort of healthy individuals injected with SARS-CoV-2 Vaccine, which will perform a longitudinal, comprehensive analysis of the SARS-CoV-2 vaccine Induced adaptive immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and aged between 18 to 59 years

Exclusion Criteria:

* High-risk epidemiology history within 14 days before enrollment
* SARS-CoV-2 specific IgG or IgM positive in serum
* Positive PCR test for SARS-CoV-2 from pharyngeal or anal swab samples
* Axillary temperature of more than 37·0°C
* Known allergy to any vaccine component
* Thyroid disease

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals to be injected with COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of anti-SARS-CoV-2 neutralizing antibody in serum | 2 years
Concentration of serum anti-SARS-CoV-2 binding antibody | 2 years
Rate of anti-SARS-CoV-2 T cell response | 2 years
The rate of SARS-CoV-2 infection | 2 years

SECONDARY OUTCOMES:
Rate of anti-SARS-CoV-2 B cell response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuxin Chen, Principal Investigator — Nanjing Drum Tower Hospital, Nanjing University Medical School; Han Shen, Principal Investigator — Nanjing Drum Tower Hospital, Nanjing University Medical School; Rui Huang, Principal Investigator — Nanjing Drum Tower Hospital, Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China